CLINICAL TRIAL: NCT05659823
Title: Impact of Guideline Recommendations for Post-caesarean Analgesia on Pain, Nausea and Pruritus
Brief Title: Postoperative Pain After Caesarian Section
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Conrad Arnfinn Bjørshol (Other Government)
Responsible Party: Sponsor-Investigator, Conrad Arnfinn Bjørshol, Senior researcher, Helse Stavanger HF
Organization: Helse Stavanger HF (Other Government)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 1399-2435
Record Dates: First submitted 2022-09-23; First posted 2022-12-21 (Actual); Last update posted 2023-04-18 (Actual); Status verified 2023-04

CONDITIONS: Pain, Postoperative; Pruritus; Nausea and Vomiting Following Administration of Anaesthetic Agent; Consumption
MeSH Terms: conditions — Pain, Postoperative; Pruritus; Nausea

STUDY DESIGN:
Intervention Model Description: Current treatment: Patients receive elective or emergency CS. Guideline recommended treatment: Only elective CS included.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Control group (Active Comparator): Elective CS patients receiving current analgesia.
  Interventions: Drug: Bupivacaine-fentanyl elective group
- Intervention group (Experimental): Elective CS patients receiving guideline recommended analgesia.
  Interventions: Drug: Bupivacaine-fentanyl-morphine elective group
- Emergency group (Experimental): Emergency CS receiving current analgesia.
  Interventions: Drug: Bupivacaine-fentanyl emergency group

INTERVENTIONS:
Drug: Bupivacaine-fentanyl-morphine elective group — Guideline recommended analgesia in elective caesarian section.
  Arms: Intervention group
Drug: Bupivacaine-fentanyl elective group — Current analgesia in elective caesarian section.
  Arms: Control group
Drug: Bupivacaine-fentanyl emergency group — Current analgesia in emergency caesarian section.
  Arms: Emergency group

SUMMARY:
To examine if perioperative pain/nausea/pruritus is altered when current standard analgesia for caesarian section (CS) is replaced with new guideline recommended analgesia.

DETAILED DESCRIPTION:
Control group (current analgesia, elective CS) is compared to current analgesia for emergency CS, and guideline recommended analgesia.

Current analgesia for CS:

Spinal hyperbaric bupivacaine 5 mg/ml, 9-11 mg. Spinal fentanyl 10-15 ug. Postoperative: Paracetamol 1g x 4, ibuprofen 400 mg x 4 po, oxycodone 10 mg (<70 kg) or 20 mg (>70 kg) x 2 po, additional oxycodone 2,5 mg iv/5 mg po when needed.

Guideline recommended analgesia for CS:

Spinal hyperbaric bupivacaine 5 mg/ml, 9-11 mg. Spinal fentanyl 12,5 ug. Spinal morphine 0,05 mg. After delivery of baby: Dexamethasone 8 mg iv, paracetamol 1g iv, parecoxib 40 mg iv.

Postoperative: Paracetamol 1g x 4, ibuprofen 600 mg x 4 po, oxycodone 2,5 mg iv/5 mg po when needed.

ELIGIBILITY:
Inclusion Criteria:

- Healthy parturient, term pregnancy, undergoing caesarian section

Exclusion Criteria:

* Patient refusal
* Maternal heart or lung disease (not including mild asthma)
* Known or suspected obstructive sleep apnoea syndrome
* Pre-eclampsia
* Body mass index > 40
* Indulin-dependent diabetes mellitus
* Contraindications to ibuprofen, dexamethasone or morphine
* Chronic pain
* Neurological disease
* Drug abuse
* Age < 18 years
* American Society of Anesthesiologists (ASA) 3
* Patients receiving other forms of anaesthesia (epidural or general)

Ages: 18 Years to 60 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 108 (Actual)
Dates: Start 2020-11-02 (Actual); Primary Completion 2021-11-05 (Actual); Study Completion 2021-11-05 (Actual)

PRIMARY OUTCOMES:
Postoperative pain at postoperative care unit arrival | Immediately upon arrival at postoperative care unit
  Postoperative pain during rest and movement measured by numeric rating scale (NRS).
Postoperative pain at 30 minutes | At postoperative care unit 30 minutes after arrival
  Postoperative pain during rest and movement measured by numeric rating scale (NRS).
Postoperative pain at 60 minutes | At postoperative care unit 60 minutes after arrival
  Postoperative pain during rest and movement measured by numeric rating scale (NRS).
Postoperative pain at 90 minutes | At postoperative care unit 90 minutes after arrival
  Postoperative pain during rest and movement measured by numeric rating scale (NRS).
Postoperative pain at 120 minutes | At postoperative care unit 120 minutes after arrival
  Postoperative pain during rest and movement measured by numeric rating scale (NRS).
Postoperative pain at maternity ward arrival | Immediately upon arrival at maternity ward
  Postoperative pain during rest and movement measured by numeric rating scale (NRS).
Postoperative pain at maternity ward 4 hours after arrival | At maternity ward 4 hours after arrival
  Postoperative pain during rest and movement measured by numeric rating scale (NRS).
Postoperative pain at maternity ward 8 hours after arrival | At maternity ward 8 hours after arrival
  Postoperative pain during rest and movement measured by numeric rating scale (NRS).
Postoperative pain at maternity ward 12 hours after arrival | At maternity ward 12 hours after arrival
  Postoperative pain during rest and movement measured by numeric rating scale (NRS).
Postoperative pain at maternity ward 16 hours after arrival | At maternity ward 16 hours after arrival
  Postoperative pain during rest and movement measured by numeric rating scale (NRS).
Postoperative pain at maternity ward 20 hours after arrival | At maternity ward 20 hours after arrival
  Postoperative pain during rest and movement measured by numeric rating scale (NRS).

SECONDARY OUTCOMES:
Postoperative nausea and vomiting at postoperative care unit | During stay at postoperative care unit, estimated average 2 hours
  Present (yes/no) during stay at the postoperative care unit
Postoperative nausea and vomiting at maternity ward | During stay at maternity ward, estimated average 22 hours
  Present (yes/no) during stay at the maternity ward
Postoperative pruritus at postoperative care unit | During stay at postoperative care unit, estimated average 2 hours
  Present (yes/no) during stay at the postoperative care unit
Postoperative pruritus at maternity ward | During stay at maternity ward, estimated average 22 hours
  Present (yes/no) during stay at the maternity ward
Postoperative additional oxycodone consumption at postoperative care unit | During stay at postoperative care unit, estimated average 2 hours
  Number of mg of oxycodone administered as additional analgetics
Postoperative additional oxycodone consumption at maternity ward | During stay at maternity ward, estimated average 22 hours
  Number of mg of oxycodone administered as additional analgetics

CONTACTS AND LOCATIONS:
Overall Officials: Conrad A Bjørshol, PhD, MD, Study Chair — Helse Stavanger HF
Locations (1):
- Stavanger University Hospital, Stavanger, Rogaland, Norway

IPD SHARING:
Plan to Share IPD: Undecided

DOCUMENTS (3):
  • Study Protocol and Statistical Analysis Plan (2022-10-03): https://cdn.clinicaltrials.gov/large-docs/23/NCT05659823/Prot_SAP_000.pdf
  • Informed Consent Form: Intervention group (2022-10-03): https://cdn.clinicaltrials.gov/large-docs/23/NCT05659823/ICF_001.pdf
  • Informed Consent Form: Informed Consent Form: Intervention group (2022-10-03): https://cdn.clinicaltrials.gov/large-docs/23/NCT05659823/ICF_002.pdf